CLINICAL TRIAL: NCT01069809
Title: A Randomized, Double-Blind, Phase 2B Study Testing the Efficacy and Safety of AGS-004 on Host Control of HIV Replication During Analytical Treatment Interruption
Brief Title: Safety and Efficacy Study of AGS-004 During Analytical Treatment Interruption
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Argos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AGS-004-003; HHSN266200600019C (Other: NIH Contract); ES-11702 (Other: DAIDS); NCT00595192 (obsolete NCT alias)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AGS-004 (Experimental): HIV-1 Immune Therapy
  Interventions: Biological: AGS-004
- Inactive Injection (Placebo Comparator): Inactive Placebo Injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AGS-004 — HIV-1 Immune Therapy
  Arms: AGS-004
Biological: Placebo — Inactive Placebo Injection
  Arms: Inactive Injection

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of AGS-004, an immune therapy, for HIV-infected individuals. Safety and effectiveness will be tested while the individuals are both taking antiretroviral therapy (ART) medication and interrupting ART medication.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and effectiveness of AGS-004, an immune therapy, for HIV-infected individuals. Safety and effectiveness will be tested while the individuals are both taking antiretroviral therapy (ART) medication and interrupting ART medication

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 to 60 years of age.
2. HIV infection.
3. Stable ART regimen for ≥ 3 months prior to Screening.
4. HIV VL level ≤ 400 copies/mL for ≥ 2 months prior to Screening.
5. HIV VL level ≤ 50 copies/mL at Screening.
6. CD4+ T cell count ≥ 450 cells/mm3 at Screening.
7. Pre-ART nadir CD4+ T cell counts ≥ 200 cells/mm³.
8. Availability of an adequate sample of frozen plasma most recently collected (no more than 90 days and preferably within 30 days) before starting ART.
9. Laboratory values within pre-defined limits at Screening and Eligibility.
10. Negative serum pregnancy test at Screening and Eligibility for females with reproductive potential, and agreement of all subjects to use a reliable form of contraception during the study and for 12 weeks after the last dose of study drug.
11. Able and willing to give adequate written informed consent, to communicate effectively with study personnel, and willing to be compliant with protocol requirements.

Exclusion Criteria:

1. HIV-2 antibody positive at Screening Visit.
2. Positive hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody (if positive HCV antibody, HCV RNA must be negative).
3. Untreated syphilis infection (positive rapid plasma reagin [RPR]).
4. Changes in ART regimen due to virologic breakthrough.
5. History of lymph node irradiation or dissection.
6. Prior use of any HIV immunotherapy or vaccine within 9 months prior to Screening.
7. Prior participation in an AGS-004 clinical study.
8. Treatment interruption of ART for > 1 month since starting the ART from which the pre-ART plasma sample was drawn.
9. Any acute infection or medical illness within 14 days prior to Screening and throughout the pre-treatment evaluation phase (Step 1).
10. Initiation of ART during the acute HIV infection stage, if date of infection known (acute infection defined as < 6 months between date of HIV infection and ART start date).
11. Pregnancy or breast-feeding.
12. Receipt of any immune modulators or suppressors within 30 days prior to Screening and throughout the pre-treatment evaluation phase (Step 1).
13. Evidence of hepatic decompensation in cirrhotic subjects: history of ascites, hepatic encephalopathy, or bleeding esophageal varices, or screening laboratory results of any of the following:

    * International Normalized Ratio (INR) of ≥ 1.5 X upper limit of normal (ULN);
    * Serum albumin < 3.3 g/dL;
    * Serum total bilirubin > 1.8 X ULN, unless history of Gilbert's disease or deemed related to treatment with atazanavir.
14. History or other clinical evidence of significant or unstable cardiac disease (e.g., angina, congestive heart failure, recent myocardial infarction, significant arrhythmia) or clinically significant electrocardiogram (ECG) abnormalities.
15. History of moderate or severe renal impairment (i.e., persistent history of creatinine clearance < 50 mL/min) or any other renal disorder deemed clinically significant by the investigator.
16. Prior history of an acquired immunodeficiency syndrome (AIDS) defining condition.
17. History or other evidence of severe illness, malignancy, immunodeficiency other than HIV, or any other condition that would make the subject unsuitable for the study in the opinion of the investigator.
18. Known allergy or sensitivity to the components of the investigational immunotherapy.
19. Active drug or alcohol use or dependence that would interfere with adherence to study requirements in the opinion of the investigator.
20. Use of systemic corticosteroids and use of topical steroids over a total area exceeding 15 cm² within 30 days prior to Screening.
21. Any investigational antiretroviral agents or use of a CCR5 inhibitor at Screening.
22. Active autoimmune disease or condition.
23. Participation in another investigational clinical study within the previous 30 days or use of investigational agents.
24. Body weight less than 30 kg.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Compare the anti-HIV effects of AGS-004 versus Placebo as measured by new HIV Viral Load setpoint after a 12 week Analytical Treatment Interruption | 38 weeks

SECONDARY OUTCOMES:
Evaluate AGS-004 versus Placebo for change in plasma HIV Viral Load levels from the value just before initiation of ART to the value at the end of the 12 week ATI. | 38 weeks
Evaluate AGS-004 versus Placebo for change from Baseline in CD4 T-Cell absolute and percentage values at Week 26 and at the end of Step 4 (for subjects continuing ATI) | 38 weeks (62 weeks for subjects continuing ATI in Step 4)
Evaluate AGS-004 versus Placebo for effects on HIV viral kinetics during the 12 week ATI, as measured my mean or median levels of plasma HIV Viral Load; assessed throughout and at the end of Step 4 (for subjects continuing ATI) | 38 weeks (62 weeks for subjects continuing ATI in Step 4)
Evaluate AGS-004 versus Placebo for change from Baseline in TEAEs, clinical laboratory evaluations, and clinical assessments. | 2 years
Evaluate AGS-004 versus Placebo for change in inflammatory markers over treatment period and ATI | 38 Weeks (62 weeks for subjects continuing ATI in Step 4)
Study immunogenicity and mechanism of action by evaluating AGS-004 versus Placebo for change from Baseline in T-cell response. | 2 years
Study immunogenicity and mechanism of action by evaluating AGS-004 versus Placebo for change from Baseline of the extent of viral evolution. | 2 years
Study immunogenicity and mechanism of action by evaluating AGS-004 versus Placebo for change from Baseline in the chromosomally integrated viral reservoir. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Jacobson, MD, Principal Investigator — Drexel University
Locations (9):
- United States (5):
  - UCDavis Research Office at CARES, Sacramento, California
  - Jacobi & North Central Bronx Hospitals, The Bronx, New York
  - AIDS Clinical Trials Unit, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Division of Infectious Disease and HIV Medicine Partnership Comprehensive Care Practice, Philadelphia, Pennsylvania
- Canada (4):
  - The Ottawa Hospital, Ottawa, Ontario
  - Clinique médicale l'Actuel, Montreal, Quebec
  - Clinique Médical du Quartier Latin, Montreal, Quebec
  - Montreal Chest Institute, Immunodeficiency Dept., Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://www.argostherapeutics.com/